CLINICAL TRIAL: NCT06507631
Title: Feasibility and Effectiveness of the Blended Care Pirate Group for Children With Unilateral Cerebral Palsy
Brief Title: Feasibility of the Blended Care Pirate Group
Status: Recruiting | Type: Observational
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Other Study IDs: 1054
Record Dates: First submitted 2024-03-06; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: Home-based rehabilitation; Constrained induced movement therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blended care pirate group: During the 8-week pirate group, children will receive two times three hour training sessions. Additionally, parents are advised to practise with their child at home for three hours per week.
  Interventions: Behavioral: Blended care pirate group

INTERVENTIONS:
Behavioral: Blended care pirate group — During the blended care pirate group, children will receive training while their less affected arm is in a sling. They will perform play-like activities with their affected arm both on-site and at home.

SUMMARY:
Rationale: In 2010 Aarts developed the pirate group in which children received constrained induced movement therapy (constrained with a sling) followed by bilateral therapy. During this pirate group children were dressed as a pirate to increase motivation and to make the sling more meaningful. This pirate group had a duration of eight weeks with three times three hour training sessions each week. However, due to COVID-19 therapists were introduced to home-based rehabilitation. Therefore they developed the blended care pirate group, which is in principle the same as the pirate group of Aarts, however one training session each week is replaced by a home-based training session. It is however not yet clear how this blended care pirate group is perceived by parents and therapists.

Objective: The aim of the current study is to investigate the feasibility and effectiveness of the blended care pirate group.

Study population: Children with unilateral cerebral palsy between 2.5 and 8 years old will participate. These children will participate in the blended care pirate group and are asked to participate in the study as well.

Intervention: The total duration of one blended care pirate group is eight weeks with two times three hour training sessions at the rehabilitation centre and additional training sessions at home. The training sessions on-site will be the same as the conventional pirate group. For the training sessions at home parents will receive instructions and material from the therapists. This intervention is developed and already planned by therapists without direct influence of the research department and can therefore be considered as standard treatment.

Main study parameters/endpoints: The primary outcome are the total training hours performed by parents at home. Additionally after the blended care pirate group parents and therapists will participate in an interview about how they perceived the blended care pirate group. Secondary outcomes are improvements in arm function during the blended care pirate group.

ELIGIBILITY:
Inclusion Criteria:

* Receiving treatment at the Sint Maartenskliniek. Care demand of parents that requires a more and better use of the affected arm and hand.
* Children with unilateral cerebral palsy
* A Manual Ability Classification System (MACS) score of I, II or III

Exclusion Criteria:

* Cognitive developmental age below 2
* Child is not able to walk independently without a walking tool

Ages: 30 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with unilateral cerebral palsy who are being reffered to the local rehabilitation centre to participate in the pirate group.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Training hours | During the 8-week intervention period
  Training hours at home will be logged by parents. The total training hours will be compared to the advised training duration of three hours per week.

SECONDARY OUTCOMES:
Interview with parents | After the 8-week intervention period
  After each pirate group, interviews with parents will be held about their experiences of training at home. A thematic analysis will be performed to analyse the interviews.
Assisting Hand Assessment (AHA) | Before and after 8-week intervention
  The AHA will be performed to measure the arm use during bimanual activities. The scale ranges between 0-100, with a higher score meaning better arm use.
Video observarion Aarts en Aarts - Determine Developmental Disregard - Revised (VOAA-DDD-R) | Before and after 8-week intervention
  The VOAA-DDD-R measures the spontaneous arm use of the affected upper limb during two activities. During one activity it is required to use both hand, and during the second it is most efficient to use both hands. The score is the difference in arm use between the two tests. This score ranges between 0-100% with a lower score indicating better spontaneous arm use.
Box and Block test (BBT) | Before and after 8-week intervention
  This test measures the unilateral gross manual dexterity. Children have to transfer blocks for one box to the other. There is no maximum score, a higher score indicating better hand function

CONTACTS AND LOCATIONS:
Overall Officials: Noël Keijsers, Prof., Principal Investigator — Donders Institute for Brain, Cognition and Behavior, Radboud University
Locations (1):
- Sint Maartenskliniek, Ubbergen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aarts PB, Jongerius PH, Geerdink YA, van Limbeek J, Geurts AC. Effectiveness of modified constraint-induced movement therapy in children with unilateral spastic cerebral palsy: a randomized controlled trial. Neurorehabil Neural Repair. 2010 Jul-Aug;24(6):509-18. doi: 10.1177/1545968309359767. Epub 2010 Apr 27. PMID 20424191